CLINICAL TRIAL: NCT00931918
Title: An Open-Label, Randomized, Phase 2 Study to Assess the Effectiveness of RCHOP With or Without VELCADE in Previously Untreated Non-Germinal Center B-Cell-like Diffuse Large B-Cell Lymphoma Patients
Brief Title: Study to Assess the Effectiveness of RCHOP With or Without VELCADE in Previously Untreated Non-Germinal Center B-Cell-like Diffuse Large B-Cell Lymphoma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C05013; U1111-1183-0186 (Registry Identifier: WHO)
Record Dates: First submitted 2009-07-01; First posted 2009-07-02 (Estimated); Results first posted 2017-01-11 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2016-11

CONDITIONS: Non-Germinal B-Cell-like (GCB) Diffuse Large B-cell Lymphoma (DLBCL)
MeSH Terms: conditions — Acromesomelic dysplasia, Maroteaux type; Lymphoma, Large B-Cell, Diffuse | interventions — Bortezomib; Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RCHOP (Active Comparator): RCHOP [rituximab, cyclophosphamide, doxorubicin, prednisone] administered as follows: rituximab 375 mg/m^2 intravenous (IV) infusion, cyclophosphamide 750 mg/m^2 IV infusion, doxorubicin 50 mg/m^2 IV injection and vincristine 1.4 mg/m^2 (maximum total dose 2 mg) IV injection on Day 1 with prednisone orally on Days 1 through 5 of a 21-day (3-week) cycle for 6 cycles.
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone
- Vc-RCHOP (Experimental): Vc-RCHOP [bortezomib (VELCADE®), rituximab, cyclophosphamide, doxorubicin, prednisone] administered as follows: bortezomib (VELCADE ®) 1.3 mg/m^2 administered intravenous (IV) push on Days 1 and 4 of each cycle with RCHOP administered as follows: rituximab 375 mg/m^2 intravenous (IV) infusion, cyclophosphamide 750 mg/m^2 IV infusion, doxorubicin 50 mg/m^2 IV injection and vincristine 1.4 mg/m^2 (maximum total dose 2 mg) IV injection on Day 1 with prednisone orally on Days 1 through 5 of a 21-day (3-week) cycle for 6 cycles.
  Interventions: Drug: Bortezomib; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone

INTERVENTIONS:
Drug: Bortezomib — Bortezomib IV
  Other Names: VELCADE®
  Arms: Vc-RCHOP
Drug: Rituximab — Rituximab IV
Drug: Cyclophosphamide — Cyclophosphamide IV
Drug: Doxorubicin — Doxorubicin IV solution
Drug: Vincristine — Vincristine IV
Drug: Prednisone — Prednisone tablet

SUMMARY:
This is a randomized, open-label, multi-center, phase 2 study of RCHOP with or without VELCADE in adult patients with previously untreated non-(Germinal B-Cell-like) GCB Diffuse Large B-cell Lymphoma (DLBCL). The study will determine whether the addition of VELCADE to RCHOP improves progression-free survival (PFS) in patients with non-GCB DLBCL.

DETAILED DESCRIPTION:
The drug tested in this study is called bortezomib (VELCADE®). VELCADE® was tested in people who have Non-Germinal Center B-Cell-like Diffuse Large B-Cell Lymphoma. This study looked at the efficacy of RCHOP [rituximab, cyclophosphamide, doxorubicin, vincristine and prednisone] with or without VELCADE®.

The study enrolled 206 patients. Participants were enrolled in one of the two open label treatment groups:

* RCHOP
* Vc-RCHOP [bortezomib (VELCADE®), rituximab, cyclophosphamide, doxorubicin, vincristine and prednisone]

Participants received treatment for up to six, 21-day cycles.

This multi-center trial was conducted in the United States. The overall time to participate in this study was up to 48 months. Participants made multiple visits to the clinic, and were followed for progression free survival and overall survival until patient withdrawal, death, or 2 years after the last participant was enrolled.

ELIGIBILITY:
Each patient must meet all of the following inclusion criteria to be enrolled in the study:

Inclusion Criteria:

* Patients with previously untreated DLBCL that has been sub classified as the non-GCB subtype.
* At least 1 measurable tumor mass.
* Availability of paraffin block with sufficient tumor tissue.
* No evidence of central nervous system lymphoma.
* Eastern Cooperative Oncology Group (ECOG) performance status of < or equal to 2.
* Female patients who are post menopausal, surgically sterile, or agree to practice 2 effective methods of contraception or abstain from heterosexual intercourse.
* Male patients who agree to practice effective barrier contraception or agree to abstain from heterosexual intercourse.

Patients meeting any of the following exclusion criteria are not to be enrolled in the study:

Exclusion Criteria:

* Diagnosed or treated for a malignancy other than DLBCL within 2 years of first dose or evidence of active malignancy other than DLBCL.
* Peripheral neuropathy of Grade 2 or greater.
* Known history of human immunodeficiency virus (HIV) infection, unless receiving highly active antiretroviral therapy (HAART).
* Active infection requiring systemic therapy.
* Major surgery within 2 weeks before first dose.
* Patients with a left ventricular ejection fraction (LVEF) or less than 45%.
* Myocardial infarction with 6 months of enrollment or evidence of current uncontrolled cardiovascular conditions as described in the protocol.
* History of allergic reaction/ hypersensitivity attributable to boron, mannitol, polysorbate 80 or sodium citrate dehydrate, or anaphylaxis or immunoglobulin E (IgE)-mediated hypersensitivity to murine proteins or to any component of rituximab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2009-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (70):
- United States (70):
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Fountain Valley Regional Hospital, Fountain Valley, California
  - St. Jude Heritage Healthcare, Fullerton, California
  - Moores Cancer Center- UCSD, La Jolla, California
  - Antelope Valley Cancer Center, Lancaster, California
  - Loma Linda University Cancer Center, Loma Linda, California
  - University of Southern California, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, Los Angeles, California
  - TORI- Central Pharmacy, Los Angeles, California
  - TORI- Central Regulatory, Los Angeles, California
  - Oncology Care Medical Associates, Montebello, California
  - Bay Area Cancer Research Group, Pleasant Hill, California
  - Wilshire Oncology Medical Group, Rancho Cucamonga, California
  - Sharp Healthcare, San Diego, California
  - Central Coast Medical Oncology Corporation, Santa Maria, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Cancer Specialists & Research Institute, Gainsville, Florida
  - Alves/ Domenech Oncology-Hematology Clinic, Hollywood, Florida
  - Florida Cancer Institute ATI, New Port Richey, Florida
  - MD Anderson Cancer Center of Orlando, Orlando, Florida
  - Coastal Oncology, PL, Ormond Beach, Florida
  - Winship Cancer Institute at Emory University, Atlanta, Georgia
  - Georgia Cancer Specialists, Atlanta, Georgia
  - Dublin Hematology and Oncology, Dublin, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Central Indiana Cancer Centers, Fishers, Indiana
  - Cancer Care Center Inc. P.C., New Albany, Indiana
  - Iowa Blood and Cancer Care, Cedar Rapids, Iowa
  - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology and Oncology Associates LLP, Sioux City, Iowa
  - Kansas City Cancer Center, LLC, Overland Park, Kansas
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - St. Agnes Hospital of Baltimore, Baltimore, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - Lahey Clinic Medical Center, Burlington, Massachusetts
  - Berkshie Hematology Oncology, Pittsfield, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Mid Michigan Physicians, Lansing, Michigan
  - Duluth Clinic, Duluth, Minnesota
  - St. Luke's Hospital Cancer Care Center, Duluth, Minnesota
  - Missouri Cancer Associates, Columbia, Missouri
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Hematology/Oncology Associates of Northern New Jersey, P.A., Morristown, New Jersey
  - Hematology Oncology Associates of South Jersey, Mount Holly, New Jersey
  - St. Luke's- Roosevelt Medical Center, New York, New York
  - Cornell, New York, New York
  - Raleigh Hematology Oncology Associates P.C., Raleigh, North Carolina
  - Summa Health System, Akron, Ohio
  - Oncology Hematology Care, Cincinnati, Ohio
  - Kaiser Group Health, Portland, Oregon
  - Hematology and Oncology Associates of NEPA, Dunmore, Pennsylvania
  - UPMC Cancer Center, Pittsburgh, Pennsylvania
  - Guthrie Clinic, Sayre, Pennsylvania
  - Berks Hematology Oncology Associates, West Reading, Pennsylvania
  - South Carolina Oncology Associates, PA, Columbia, South Carolina
  - Chattanooga Oncology and Hematology Associates, PC, Chattanooga, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - Texas Oncology Cancer Center, Austin, Texas
  - US Oncology- Central Drug, Fort Worth, Texas
  - US Oncology- Central Laboratory, Fort Worth, Texas
  - Oncology Consultants P.A., Houston, Texas
  - Oncology Consultants, Houston, Texas
  - US Oncology- Central Regulatory, The Woodlands, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Texoma Cancer Center, Wichita Falls, Texas
  - Virginia Cancer Institute, Richmond, Virginia
  - Puget Sound Cancer Centers, Edmonds, Washington
  - Northwest Cancer Specialists PC, Vancover, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 69 investigative sites in the United States from 13 October 2009 to 15 August 2015.
Pre-assignment Details: Participants with a diagnosis of Non-Germinal Center B-Cell-like Diffuse Large B-Cell Lymphoma were enrolled equally in 1 of 2 treatment groups: RCHOP [rituximab, cyclophosphamide, doxorubicin, prednisone] or Vc-RCHOP [bortezomib (VELCADE®), rituximab, cyclophosphamide, doxorubicin, prednisone] for 6, 21 day cycles.
Period: Overall Study
Arm/Group | RCHOP | Vc-RCHOP
Started | 103 | 103
Safety Population: Received Study Drug | 100 | 101
Completed | 86 (Completed the maximum of 6 cycles.) | 86 (Completed the maximum of 6 cycles.)
Not Completed | 17 | 17
Not completed — Adverse Event | 4 | 6
Not completed — Progressive Disease | 2 | 1
Not completed — Symptomatic Deterioration | 1 | 0
Not completed — Withdrawal by Patient | 3 | 4
Not completed — Other Reason not Specified | 4 | 4
Not completed — Did not receive study drug | 3 | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) Population included all randomized participants who had at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | RCHOP | Vc-RCHOP | Total
Number analyzed (Participants) | 100 | 101 | 201
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (14.60) | 61.9 (13.81) | 60.9 (14.21)
Age, Customized [Number; unit: participants]
  ≤ 65 years | 58 | 55 | 113
  > 65 years | 42 | 46 | 88
Gender [Count of Participants; unit: Participants]
  Female | 43 | 51 | 94
  Male | 57 | 50 | 107
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 14 | 20
  Not Hispanic or Latino | 90 | 82 | 172
  Unknown or Not Reported | 4 | 5 | 9
Race/Ethnicity, Customized [Number; unit: participants]
  White | 77 | 79 | 156
  Black or African American | 10 | 9 | 19
  Asian | 6 | 5 | 11
  Other | 4 | 5 | 9
  Not Reported | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 100 | 101 | 201
Height [Mean (Standard Deviation); unit: cm] — Height data is available for n=99, 99 participants, respectively.
  cm | 171.1 (11.30) | 170.3 (11.48) | 170.7 (11.37)
Weight [Mean (Standard Deviation); unit: kg] | 85.19 (20.684) | 82.86 (21.745) | 84.02 (21.203)
Body Surface Area [Mean (Standard Deviation); unit: m^2] — Body Surface Area (m²) is calculated based on patient's height and weight, and is defined as ([Height(cm) x Weight (kg)]/3600). Body Surface Area data is available for n=99, 99 participants respectively.
  m^2 | 2.002 (0.2830) | 1.970 (0.3040) | 1.986 (0.2934)

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) in Patients With Non-germinal Center B-cell-like (Non-GCB) Diffuse Large B-cell Lymphoma (DLBCL)
Description: PFS is defined as the time in months from the date of randomization to the date of first documentation of progressive disease (PD) or death from any cause. The date of progression is the earliest date of a computed tomography/positron emission tomography (CT/PET) scan that shows evidence of PD. For a participant that has not progressed and is alive at the end of his/her study follow-up or at the time of start of an alternate therapy (whichever is first), PFS is censored at the last overall response assessment that is stable disease or better, and which is prior to the start of the alternate therapy, if any. Disease response was assessed using International Working Group (IWG)-revised response criteria for malignant lymphoma. PD= any new lesion or increase by > 50% of previously involved sites from nadir.
Time Frame: Median Follow-up of 34.3 months for RCHOP arm and 34.4 months for Vc-RCHOP arm
Population: Modified Intent-to-treat (mITT) Population included all randomized participants who received study drug and who had a central laboratory-confirmed Non-Germinal Center B-Cell (non-GCB) subtype.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | RCHOP | Vc-RCHOP
Number analyzed (Participants) | 91 | 92
months | NA [NA to NA] — Median not estimable due to the low number of participants with events. | NA [NA to NA] — Median not estimable due to the low number of participants with events.

2. Primary Outcome: Progression-Free Survival Rate
Description: PFS is defined as the time in months from the date of randomization to the date of first documentation of progressive disease (PD) or death from any cause. The date of progression is the earliest date of a computed tomography/positron emission tomography (CT/PET) scan that shows evidence of PD. For a participant that has not progressed and is alive at the end of his/her study follow-up or at the time of start of an alternate therapy (whichever is first), PFS is censored at the last overall response assessment that is stable disease or better, and which is prior to the start of the alternate therapy, if any. Disease response was assessed using International Working Group (IWG)-revised response criteria for malignant lymphoma. PD= any new lesion or increase by > 50% of previously involved sites from nadir. The progression-free survival rate is defined as the Kaplan-Meier (KM) estimate of progression-free survival at 2 years.
Time Frame: 2 Years (Median Follow-up of 34.3 months for RCHOP arm and 34.4 months for Vc-RCHOP arm)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | RCHOP | Vc-RCHOP
Number analyzed (Participants) | 91 | 92
percentage of participants | 78 | 82

3. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from the date of randomization to the date of death from any cause. A participant who is alive at the end of his/her study follow-up is censored at the date of last contact.
Time Frame: Median Follow-up of 34.3 months for RCHOP arm and 34.4 months for Vc-RCHOP arm
Population: MITT Population included all randomized participants who received study drug and who had a central laboratory-confirmed Non-Germinal Center B-Cell (non-GCB) subtype.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | RCHOP | Vc-RCHOP
Number analyzed (Participants) | 91 | 92
months | NA [NA to NA] — Median not estimable due to the low number of participants with events. | NA [NA to NA] — Median not estimable due to the low number of participants with events.

4. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants with the best overall response complete response (CR) + partial response (PR). Disease response was assessed using International Working Group (IWG)-revised response criteria for malignant lymphoma. CR=disappearance of all evidence of disease and PR=regression of measurable disease and no new sites.
Time Frame: End of Cycle 2, End of Treatment (Cycle 6) [Median of 16 weeks on treatment]
Population: Response-Evaluable Population included all randomized participants who had at least 1 dose of study drug, who had a central laboratory-confirmed non-GCB subtype with measurable disease at Baseline and at least 1 post-baseline response assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RCHOP | Vc-RCHOP
Number analyzed (Participants) | 86 | 90
percentage of participants
  End of Cycle 2 | 93 [86 to 97] | 90 [82 to 95]
  End of Treatment (Cycle 6) | 88 [80 to 94] | 84 [76 to 91]
  Best Overall Response Rate | 98 [92 to 99] | 96 [89 to 98]

5. Secondary Outcome: Complete Response Rate
Description: Complete Response Rate is defined as the percentage of participants with the best response of Complete Response (CR). Disease response was assessed using International Working Group (IWG)-revised response criteria for malignant lymphoma. CR=Disappearance of all evidence of disease.
Time Frame: End of Cycle 2, End of Treatment (Cycle 6) [Median of 16 weeks on treatment]
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RCHOP | Vc-RCHOP
Number analyzed (Participants) | 86 | 90
percentage of participants
  End of Cycle 2 | 23 [16 to 33] | 16 [9 to 24]
  End of Treatment (Cycle 6) | 45 [35 to 56] | 56 [45 to 65]
  Best Complete Response Rate | 49 [39 to 59] | 56 [45 to 65]

6. Secondary Outcome: Duration of Response
Description: Duration of response is defined as the time (in months) from the date of first documentation of confirmed complete response (CR) or partial response (PR) to the date of first documentation of progressive disease (PD), relapse from CR or death related to disease. For a participant who has not progressed and is not known to have died due to disease under study at the end of his/her study follow-up or at the time of start of an alternate therapy (whichever is first), duration of response is censored at the last overall response assessment that is stable disease or better, and which is prior to the start of the alternate therapy, if any. Disease response was assessed using IWG-revised response criteria for malignant lymphoma. CR=Disappearance of all evidence of disease and PR=Regression of measurable disease and no new sites and PD= any new lesion or increase by > 50% of previously involved sites from nadir.
Time Frame: Median Follow-up of 34.3 months for RCHOP arm and 34.4 months for Vc-RCHOP arm
Population: Participants from the Response-Evaluable Population included all randomized participants who had at least 1 dose of study drug, who had a central laboratory-confirmed non-GCB subtype with measurable disease at Baseline and at least 1 post-baseline response assessment who had a CR or PR
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | RCHOP | Vc-RCHOP
Number analyzed (Participants) | 84 | 86
months | NA [NA to NA] — Median not estimable due to the low number of participants with events. | NA [NA to NA] — Median not estimable due to the low number of participants with events.

7. Secondary Outcome: Fluorodeoxyglucose Positron Emission Tomography (FDG-PET) Negative Rate
Description: FDG-PET negative rate is defined as the percentage of participants FDG-PET negative at the given time-point.
Time Frame: End of Cycle 2 and End of Treatment (Cycle 6) [Median of 16 weeks on treatment]
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RCHOP | Vc-RCHOP
Number analyzed (Participants) | 86 | 90
percentage of participants
  End of Cycle 2 | 42 [32 to 52] | 37 [27 to 47]
  End of Treatment (Cycle 6) | 53 [43 to 64] | 59 [49 to 68]

8. Secondary Outcome: Time to Progression (TTP)
Description: TTP is defined as the time from the date of randomization to the date of first documentation of progressive disease, relapse from CR, or death related to disease under study if participant did not have any documentation of disease progression prior to death caused by lymphoma or complications thereof. For a participant who has not progressed and is not known to have died due to disease under study at the end of his/her study follow-up or at the time of start of an alternate therapy (whichever is first), TTP is censored at the last overall response assessment that is stable disease or better, and which is prior to the start of the alternate therapy, if any. Disease response was assessed using International Working Group (IWG)-revised response criteria for malignant lymphoma. PD= any new lesion or increase by > 50% of previously involved sites from nadir.
Time Frame: Median Follow-up of 34.3 months for RCHOP arm and 34.4 months for Vc-RCHOP arm
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | RCHOP | Vc-RCHOP
Number analyzed (Participants) | 91 | 92
months | NA [NA to NA] — Median is not estimable due to the low number of participant with events. | NA [NA to NA] — Median is not estimable due to the low number of participant with events.

9. Secondary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (TEAEs) by Category
Description: Percentage of participants in the following categories: • At least 1 TEAE • Drug-related, TEAEs • Grade 3 or higher TEAEs. Grade 3 are AEs of Severe Intensity • Grade 3 or higher drug-related, TEAEs • TEAEs resulting in study drug discontinuation • Serious TEAEs An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug. A Serious Adverse Event (SAE) is any experience that suggests a significant hazard, contraindication, side effect or precaution that: results in death, is life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant.
Time Frame: First dose of study drug through 30 days after the last dose of study drug (Up to 26 Weeks)
Population: Safety Population included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | RCHOP | Vc-RCHOP
Number analyzed (Participants) | 100 | 101
percentage of participants
  At Least 1 TEAE | 100 | 99
  Drug-related, TEAEs | 88 | 95
  Grade 3 or higher TEAEs | 71 | 79
  Grade 3 or Higher Drug-related, TEAEs | 55 | 68
  TEAEs Resulting in Study Drug Discontinuation | 4 | 6
  Serious TEAEs | 31 | 34

10. Secondary Outcome: Percentage of Participants With Chemistry and Hematology Laboratory Values Grade 3 or Higher
Description: Percentage of participants who shifted from a National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Grade 0, 1, or 2 at Baseline to a Grade 3 or higher on study (worst post-baseline grade). Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe or medically significant but not immediately life-threatening, Grade 4=Life-threatening consequences and 5=Death related to AE.
Time Frame: Days 1, 4 and 10 of each cycle and end of treatment visit (Median of 16 weeks on treatment)
Population: Safety Population included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | RCHOP | Vc-RCHOP
Number analyzed (Participants) | 100 | 101
percentage of participants
  Lymphocytes | 70 | 86
  WBC Count | 68 | 69
  Neutrophils | 65 | 70
  Platelets | 18 | 39
  Hemoglobin | 10 | 15
  Hyperglycemia | 14 | 9
  Hypokalemia | 13 | 14
  Hypophosphatemia | 7 | 10
  Hyponatremia | 4 | 3
  Alanine aminotransferase (ALT) increased | 2 | 1
  Aspartate aminotransferase (AST) increased | 1 | 2

ADVERSE EVENTS:
Time Frame: First dose of study drug through 30 days after the last dose of study drug (Up to 26 Weeks)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | RCHOP | Vc-RCHOP
Serious Adverse Events (participants affected / at risk) | 31/100 | 34/101
Other Adverse Events (participants affected / at risk) | 100/100 | 100/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RCHOP (N=100) | Vc-RCHOP (N=101)
Febrile neutropenia (Blood and lymphatic system disorders) | 8 | 7
Neutropenia (Blood and lymphatic system disorders) | 5 | 1
Pancytopenia (Blood and lymphatic system disorders) | 2 | 1
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Leukopenia (Blood and lymphatic system disorders) | 2 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Herpes zoster (Infections and infestations) | 1 | 3
Pneumonia (Infections and infestations) | 3 | 1
Sepsis (Infections and infestations) | 1 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0 — One treatment-emergent death of septic shock occurred during treatment with RCHOP and is considered related to study treatment by the investigator.
Gastroenteritis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 1 | 0
Cellulitis staphylococcal (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Pyrexia (General disorders) | 4 | 4
Asthenia (General disorders) | 1 | 2
Fatigue (General disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 6
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Vomiting (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Duodenal obstruction (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Melaena (Gastrointestinal disorders) | 0 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 4
Metabolic encephalopathy (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0
Angina unstable (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 — One treatment-emergent death, Cardio-respiratory arrest occurred during treatment with Vc-RCHOP considered related to study treatment by investigator (other SAEs dehydration,febrile neutropenia,intestinal obstruction,acute kidney injury and syncope).
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 3
Hypotension (Vascular disorders) | 0 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 1
Nuclear magnetic resonance imaging abnormal (Investigations) | 1 | 0
Transaminases increased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Troponin increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 1
Fluid replacement (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RCHOP (N=100) | Vc-RCHOP (N=101)
Anaemia (Blood and lymphatic system disorders) | 30 | 37
Leukopenia (Blood and lymphatic system disorders) | 21 | 13
Lymphopenia (Blood and lymphatic system disorders) | 8 | 6
Neutropenia (Blood and lymphatic system disorders) | 44 | 38
Thrombocytopenia (Blood and lymphatic system disorders) | 20 | 39
Tachycardia (Cardiac disorders) | 5 | 4
Lacrimation increased (Eye disorders) | 6 | 2
Vision blurred (Eye disorders) | 5 | 7
Abdominal distension (Gastrointestinal disorders) | 3 | 9
Abdominal pain (Gastrointestinal disorders) | 9 | 11
Constipation (Gastrointestinal disorders) | 45 | 44
Diarrhoea (Gastrointestinal disorders) | 26 | 27
Dry mouth (Gastrointestinal disorders) | 7 | 4
Dyspepsia (Gastrointestinal disorders) | 13 | 10
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 | 6
Nausea (Gastrointestinal disorders) | 56 | 51
Oral pain (Gastrointestinal disorders) | 6 | 0
Stomatitis (Gastrointestinal disorders) | 24 | 19
Vomiting (Gastrointestinal disorders) | 18 | 19
Asthenia (General disorders) | 8 | 7
Chills (General disorders) | 9 | 6
Fatigue (General disorders) | 70 | 55
Oedema peripheral (General disorders) | 14 | 25
Pain (General disorders) | 8 | 2
Pyrexia (General disorders) | 14 | 11
Herpes zoster (Infections and infestations) | 2 | 10
Oral candidiasis (Infections and infestations) | 6 | 4
Upper respiratory tract infection (Infections and infestations) | 8 | 6
Urinary tract infection (Infections and infestations) | 7 | 8
Infusion related reaction (Injury, poisoning and procedural complications) | 5 | 9
Alanine aminotransferase increased (Investigations) | 6 | 4
Aspartate aminotransferase increased (Investigations) | 6 | 8
Haemoglobin decreased (Investigations) | 5 | 8
Neutrophil count decreased (Investigations) | 13 | 19
Platelet count decreased (Investigations) | 11 | 12
Weight decreased (Investigations) | 10 | 9
Weight increased (Investigations) | 2 | 6
White blood cell count decreased (Investigations) | 10 | 18
Decreased appetite (Metabolism and nutrition disorders) | 27 | 24
Dehydration (Metabolism and nutrition disorders) | 14 | 17
Hyperglycaemia (Metabolism and nutrition disorders) | 8 | 13
Hypocalcaemia (Metabolism and nutrition disorders) | 5 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 18 | 20
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 | 7
Hyponatraemia (Metabolism and nutrition disorders) | 7 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 5 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 11
Bone pain (Musculoskeletal and connective tissue disorders) | 6 | 13
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 8 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 10 | 8
Neck pain (Musculoskeletal and connective tissue disorders) | 6 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 7
Dizziness (Nervous system disorders) | 17 | 15
Dysgeusia (Nervous system disorders) | 21 | 17
Headache (Nervous system disorders) | 23 | 18
Memory impairment (Nervous system disorders) | 5 | 1
Neuropathy peripheral (Nervous system disorders) | 20 | 32
Paraesthesia (Nervous system disorders) | 2 | 7
Peripheral sensory neuropathy (Nervous system disorders) | 23 | 21
Anxiety (Psychiatric disorders) | 10 | 10
Insomnia (Psychiatric disorders) | 26 | 29
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 | 10
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 12 | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 7 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 51 | 44
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 3
Rash (Skin and subcutaneous tissue disorders) | 12 | 4
Hypotension (Vascular disorders) | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.